



## STATISTICAL ANALYSIS PLAN

# AN OPEN LABEL, SINGLE ARM, SINGLE CENTER CLINICAL STUDY IN HEALTHY SUBJECTS TO QUALIFY AN IN-HOUSE REFERENCE STANDARD BATCH OF SCI-B-VAC $^{\rm TM}$

Protocol Number: SciB018

Protocol Version 3.0 amendment #2 dated 01-05-2016

SAP Final Version 4.0: 25-May-2017







Medicine Stat

| 1. | ABE | BREVIATIONS | 4 |
|----|------|-------------------------------------------|-----|
| 2. | INT | RODUCTION | . 6 |
| : | 2.1 | Objectives | . 6 |
| ; | 2.2 | Design | 6 |
| 2 | 2.3 | Study Flow-chart | 8 |
| : | 2.4 | Study Populations | 10 |
| 2 | 2.5 | Study Endpoints | 10 |
| 2 | 2.6 | Sample size | 11 |
| : | 2.7 | Interim Analyses | 12 |
| | 2.8 | Final Analyses | 12 |
| 3. | Stat | istical methods | 12 |
| ; | 3.1 | General | 12 |
| ; | 3.2 | Data Summaries | 12 |
| ; | 3.3 | Continuous | 12 |
| ; | 3.4 | Categorical | 14 |
| ; | 3.5 | Protocol Deviations | 14 |
| 4. | Ana | lysis Plan | 14 |
| | 4.1 | Introduction | 14 |
| 4 | 4.1 | Disposition of Subjects | 14 |
| 4 | 4.2 | Demographics and Baseline Characteristics | 14 |
| 4 | 4.3 | Compliance | 15 |
| 4 | 4.4 | Primary Endpoint Analysis | 15 |
| • | 4.5 | Secondary Endpoints Analysis | 16 |
| | 4.6 | Exploratory Endpoints Analysis | 16 |



Version 4.0 25-May-2017

| 4 | 4.7 | Safety analysis | . 16 |
|---|---|---|---|
| 5. | Арр | endix I: TABLES TO BE INCLUDED IN THE statistical REPORT | . 20 |
| 6. | APF | PENDIX II: LISTINGS TO BE INCLUDED IN THE statistical REPORT | . 22 |
| 7. | APF | PENDIX III: figures | . 23 |
| 8. | APF | PENDIX IV: listings of Screening Failures | . 24 |
| 9. | vers | sion History: | . 25 |
| 10 | . App | roval for implementation of | . 26 |




#### 1. ABBREVIATIONS

Abbreviation/Term Definition

AE Adverse Events

ANA Antinuclear antibodies

ALT Alanine transaminase

Anti-HBc Antibodies to hepatitis B core antigen

Anti-HBs Antibodies to HBsAg

Anti-HCV Antibodies to hepatitis C virus AST Aspartate aminotransferase

BMI Body Mass Index
BP Blood Pressure
BUN Blood Urea Nitrogen
CBC Complete Blood Count

cm Centimeter

CRC Clinical Research Center

CRF Case Report Form ECG Electrocardiogram

FDA Food and Drug Administration

GCP Good Clinical Practice

GGT Gamma glutamyl transferase
GLP Good Laboratory Practice
GMP Good Manufacturing Practice

GMR Geometric mean ratio
GSK Glaxo Smith Kline

h Hours

HbsAg Hepatitis B Surface Antigen HIV Human immunodeficiency virus

HR Heart Rate

ICF Informed Consent Form

ICH International Conference on Harmonization

IEC Independent Ethics Committee

IM Intramuscular

IMP Investigational Medicinal Product

IRB Institutional Review Board

Kg Kilogram Meter

MedDra Medical Dictionary for Regulatory Activities

mg Milligram min Minute

mITT Modified intention-to-treat analysis

ml Milliliter

MOH Ministry of Health
N/A Not Applicable
°C Degrees centigrade
PI Principal Investigator

PT Prothrombin Time PT Preferred Term






PT/INR Prothrombin time/International Normalized Ratio

QA Quality Assurance

R&D Research and Development

RBC Red blood cells

RDW RBC distribution width

RR Respiration rate

SAS Statistical Analysis Software SAE Serious Adverse Event SOC System Organ Class

SOP Standard Operation Procedures

SPR Seroprotection rate

SUSAR Suspected unexpected serious adverse reaction

TASMC Tel Aviv Sourasky Medical Center
TEAE Treatment emergent adverse events

WBC White blood cell

WHO World Health Organization

μg Microgram



#### 2. INTRODUCTION

## 2.1 Objectives

This document details the statistical analysis that will be performed for the SciVac Ltd. Phase IV study SciB018.

The study primary objective is:

 To validate the new in-house reference standard vaccine for routine quality control purposes, in compliance with the European Pharmacopeia and the Israeli Ministry of Health.

The secondary objectives are:

- To characterize the immunological response throughout the study.
- To monitor the subjects for safety throughout the study period

The Exploratory Objectives are:

- To collect blood samples for the in vitro validation of anti-HBs, anti-preS1 and anti-preS2 antibodies assays.
- To assess the anti-preS1 and anti-preS2 antibodies responses upon vaccination.
- To investigate additional protective mechanisms of action and the type of immune response triggered by the vaccination. No genetic tests will be performed.

#### 2.2 Design

This will be a post-marketing, open-label, single arm study in healthy volunteers who had never been vaccinated with any hepatitis B vaccine and who are HBs antigen, anti-HBc and anti-HBsAg antibodies seronegative.

The study assessments will be performed as described in the study flow chart (See section 2.3).

This study will consist of three periods:

#### Screening Period (Visit 1: up to 1 month prior to first vaccination)

After signing of the informed consent form (ICF), screening procedures will be carried out as specified in the study protocol.

## Treatment and Follow-up Period (Visits 2-8: Months 0-6)

Subject identification number will be assigned to all eligible subjects following assessment of inclusion and exclusion criteria.




All eligible subjects will receive Sci-B-Vac<sup>TM</sup> vaccine. The treatment phase will include three I.M. doses of Sci-B-Vac<sup>TM</sup> administered in the deltoid muscle on Month 0, Month 1, and Month 6. Subjects will be followed up for safety evaluations and for efficacy (by anti-HBs, anti-pre-S1 and anti-pre-S2 testing), every month. The previous injection site will be inspected before the second and third administration.

The following assessments will be performed during each treatment visit: recording of AEs and concomitant medications, vital signs and blood tests for quantitative anti-HBs, anti-preS1 and anti-preS2 antibodies and safety assessment (including blood and urine laboratory tests). Female subjects will also undergo a urine pregnancy before each injection. Vital signs are not required on follow-up visits when vaccine is not administered.

## Post-Vaccination Follow-up Period (Visits 9-11: Months 7, 9 and 12)

Additional subject follow-up visits will take place 1, 3 and 6 months after the last vaccine administration. On each visit, subjects will be inquired about AEs and concomitant medications, and blood samples for quantitative anti-HBs, anti-preS1 and anti-preS2 antibodies levels will be drawn. The last visit (Month 12) is a study termination visit in which all subjects will also undergo physical examination, laboratory safety assessments (CBC, blood chemistry and urinalysis), vital signs measurement and a 12-lead ECG. In addition, female subjects will undergo a urine pregnancy test.




# 2.3 Study Flow-chart

| Visit Number | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit Name | Screening | Treatment | Treatment | Follow- | Follow- | Follow- | Follow- | Treatment | Follow- | Follow- | Study |
| Visit Ivalle | | 1 | 2 | up | up | up | up | 3 | up | up | Termination |
| Month (Week) of the | -1 ((-)4) - | $\theta$ ( $\theta^1$ ) | $1(4^1)$ | $2(8^{1})$ | $3(12^1)$ | $4(16^1)$ | $5(20^{1})$ | 6(241() | 7(281) | 9(36²) | $12(48^2)$ |
| Study | 0 | | | | | | | | | | |
| Activity | | | | | | | | | | | |
| ICF | X | | | | | | | | | | |
| Demographics | X | | | | | | | | | | |
| Inclusion/Exclusion | X | X | | | | | | | | | |
| Medical history | X | | | | | | | | | | |
| Vital signs <sup>3</sup> | X | $X^4$ | $X^4$ | | | | | $X^4$ | | | X |
| Smoking status | X | | | | | | | | | | |
| Weight, height, BMI | X | | | | | | | | | | |
| Physical examination | X | | | | | | | | | | X |
| Blood safety tests <sup>5</sup> | X | X <sup>6</sup> | X <sup>6</sup> | | | | | X <sup>6</sup> | | | X |
| Screening serology <sup>7</sup> | X <sup>8</sup> | | | | | | | | | | |
| General urinalysis | X | X <sup>6</sup> | X <sup>6</sup> | | | | | X <sup>6</sup> | | | X |
| Serum β-HCG | X | | | | | | | | | | |
| Urine pregnancy test | | X <sup>6</sup> | X <sup>6</sup> | | | | | X <sup>6</sup> | | | X |
| 12-lead ECG | X | | | | | | | | | | X |
| Sci-B-Vac™ injection <sup>9</sup> | | X | X | | | | | X | | | |
| Local reaction grading | | $X^{14}$ | X <sup>14, 15</sup> | $X^{15}$ | | | | $X^{14}$ | $X^{15}$ | | |
| Serologic markers for | X <sup>8,10</sup> | $X^{6,11}$ | X <sup>6,11</sup> | $X^{11}$ | X <sup>11</sup> | X <sup>11</sup> | X <sup>11</sup> | X <sup>6, 11</sup> | $X^{11}$ | X <sup>11</sup> | $X^{12}$ |
| hepatitis B infection | | | | | | | | | | | |
| Serologic response to immunization 13 | | X <sup>6</sup> | X <sup>6</sup> | X | X | X | X | X <sup>6</sup> | X | X | X |
| immunization <sup>13</sup> | | | | | | | | | | | |
| Sample for further | | X <sup>6</sup> | X <sup>6</sup> | X | X | X | X | X <sup>6</sup> | X | X | X |
| investigations | | | | | | | | | | | |
| Adverse Events | Recorded throughout the study | | | | | | | | | | |
| Concomitant Medications | | | | | Recor | ded througho | out the study | | | | |




- 1 ± 3 days (Visit2/Treatment 1 may be performed up to 4 weeks +3 days from screening visit)
- $2 \pm 8$  days
- 3 Sitting BP, HR, RR, oral temperature
- 4 Within 60 min before vaccine administration and at 60 ( $\pm$  15) min after vaccination
- 5 CBC, blood chemistry, PT/INR (screening only) see Appendix B
- <sup>6</sup> Prior to vaccine administration
- <sup>7</sup> Anti HIV (Ab type 1&2), anti-HCV Ab, anti-HAV IgM antibodies, ANA (See Appendix B)
- 8 Positive serology excludes from participation in the study
- 9 One IM injections of 1.0 ml into the deltoid muscle. The previous injection site will be inspected before the second and third administration. Subjects will remain for
- observation in the CRC for at least 1 hour after injections.
- 10 HBsAg, anti-HBs antibodies (also markers for previous vaccination), total anti-HBc antibodies and IgM anti-HBc antibodies.
- 11 HBsAg only.
- 12 HBsAg, Total anti-HBc antibodies and IgM anti-HBc antibodies
- 13 Anti-HBsAg, anti-preS1 and anti-preS2 antibodies
- $^{14}$  Local reaction grading after vaccination
- 15 Local reaction grading of previous vaccine administration and follow up until symptoms resolve



Statistical Analysis Plan

# 2.4 Study Populations

Up to ninety two (92) healthy subjects will be enrolled in the study

Intent-to-Treat (ITT) Population includes all enrolled subjects who were vaccinated at least once with Sci-B-Vac<sup>™</sup>. The Safety population will be same as ITT population.

Modified Intent-to-Treat (mITT) population is a subset of the ITT set. This set will consist of all enrolled subjects who were vaccinated at least once with Sci-B-Vac<sup>™</sup> and had at least one post vaccination follow-up visit, fully comply with the study protocol, had no violation of any of the inclusion/exclusion criteria and did not demonstrate an anamnestic response after the 1<sub>st</sub> administration of Sci-B-Vac. An anamnestic response revealed by Sci-B-Vac is defined as anti-HBs level above 6000mIU/mI (the highest titer recorded upon Sci-B-Vac 1<sub>st</sub> injection) in a subject with no detectable anti-HBs antibody at visits 1 and 2. Subjects who early terminated the study but reached the primary endpoint will be included as well. Subjects who did not complete the full-course of vaccination (i.e. 3 injections) and did not reach SPR will be excluded from the mITT set. This analysis set will serve as the primary analysis set for efficacy and safety inference.

**Full Treatment (FT) set** is a subset of the mITT analysis set and will consist of all subjects who were vaccinated 3 times with Sci-B-Vac<sup>™</sup> and had at least one visit following the 3rd vaccination.

## 2.5 Study Endpoints

## **Primary Endpoint:**

Seroprotection rate (SPR), defined as the proportion of subjects with anti-HBs antibody titer at least equal to 10mIU/mI, at Month 7 (i.e. one month after the third immunization with Sci–B-Vac<sup>TM</sup>). Subjects early terminated from the study for any reason at any time while having an anti-HBs antibody concentrations  $\geq 10\text{mIU/mI}$  will be considered among those who met endpoint.

#### Secondary Endpoints:

- 1. SPR one month after the first injection and at every month until Month 6 inclusive and at months 9 and 12.
- 2. Percentage of subjects with anti-HBs antibodies titer ≥ 100mIU/ml at one month after the first injection and then at every month until Month 7 inclusive and at months 9 and 12.
- 3. The geometric mean concentration (GMC) as determined by anti-HBsAg antibody titers at Month 0, then at every month until Month 7 inclusive and at months 9 and 12.






# **Exploratory Endpoints:**

- 1. The anti-preS1 antibody titers measured at Month 0, then at every month until Month 7 inclusive and at months 9 and 12.
- 2. The anti-preS2 antibody titers measured at Month 0, then at every month until Month 7 inclusive and at months 9 and 12.

## 2.6 Sample size

Sample size determination was performed under the following assumptions:

- The primary endpoint for the study is the Seroprotection Rate (SPR), defined as the proportion of subjects with anti-HBs antibody titer at least equal to 10mIU/mI, at Month 7 (i.e. one month after the third immunization with Sci-B-Vac<sup>™</sup>). Subjects early terminated from the study for any reason at any time while having an anti-HBs antibody concentrations ≥ 10mIU/mI will be considered among those who met endpoint.
- It is expected that the true rate of SPR following treatment with Sci–B-Vac<sup>™</sup> is 95% or more.
- The principal analysis of the primary endpoint will be a non-inferiority analysis testing the below hypothesis:

H0: P-p0 ≤ -Margin

H1: P-p0 > -Margin

- Where p0, the assumed true SPR is 95% and the non-inferiority margin is 9.0%, employing that study will be considered successful if the lower bound of the 95.0% exact CI will be 86.0% or more (lower non-inferiority limit).
- The rationale for sample size calculation is based on demonstrating an expected SPR rate of 95%. The lower bound of a calculated 95% confidence interval (CI) using Exact binomial method ensures that the actual SPR rate will not exceed the calculated lower limit (will not be lower than the lower bound).
- The sample size is adjusted to a total of 94 subjects to account for an anticipated withdrawal rate of approximately 20%.
- The sample size was enlarged to 92, to ensure sufficient sample size is achieved upon the exclusion of isolated case of anamnestic response. An anamnestic response revealed by Sci-B-Vac is defined as anti-HBs level above 6000mIU/ml (the highest titer recorder upon Sci-B-Vac 1st injection in naïve subject) in eligible subject with no detectable anti-HBs antibody at visits 1 and 2.

## Sample Size Justification:




When the sample size is 70, a one-sided 95.0% confidence interval (CI) for a single proportion using Exact binomial method will demonstrate a lower bound of 86.0% or more for an expected proportion of 0.95.

## 2.7 Interim Analyses

The percent of subjects who achieved the primary endpoint will be tested at various time points. As soon as approximately 95% of the subjects (from at least 50 subjects) will be found seroprotected (having anti-HBs antibody concentrations ≥ 10mIU/mI) then the primary efficacy endpoint will be achieved and the analysis will be considered a formal interim analysis and will be reported. A second interim analysis will be performed after all subjects have completed all three injections. Subjects who early terminated the study but reached the primary endpoint prior to termination will be included in the analysis.

Interim analysis reports will include all efficacy and safety information collected up to the interim analysis cut-off date. Exploratory endpoints (anti-pre-S1 and anti-pre-S2 testing) will not be included in the interim reports.

## 2.8 Final Analyses

The final analysis will include all the subjects who completed 12 months of follow-up, fully comply with the study protocol and have no inclusion/exclusion criteria violation. Subjects who early terminated the study but achieved the primary endpoint prior to withdrawal will be included as well (mITT population). If 95% of the subjects will be found seroprotected (having anti-HBs antibody concentrations ≥ 10mIU/mI) then the primary endpoint will be achieved.

## 3. STATISTICAL METHODS

#### 3.1 General

The overall significance level for this study will be 5% using two-tailed tests.

The data will be analysed using the SAS ® version 9.3 or higher (SAS Institute, Cary North Carolina).

#### 3.2 Data Summaries

All measured variables and derived parameters will be listed individually and, if appropriate, tabulated by descriptive statistics.

## 3.3 Continuous

For continuous variables summary tables will be provided giving sample size, arithmetic mean, standard deviation, standard error, median, minimum and maximum and 95% confidence interval for means (id appropriate). Summary statistics of Anti-HBs antibody concentrations






and Anti-PreS1 and Anti-PreS2 antibodies concentrations will use geometric means due to the expected dispersion and skewness of the data.




## 3.4 Categorical

For categorical variables summary tables will be provided giving sample size, absolute and relative frequency.

#### 3.5 Protocol Deviations

Listing of protocol deviations will be provided.

#### 4. ANALYSIS PLAN

#### 4.1 Introduction

All summaries and analyses documented below will be presented in the final integrated statistical/clinical report and tables that will be based on the E3 guidelines published by ICH. However, it is noted here that no analysis plan prepared in advance of database lock can be absolutely definitive and so the final report may contain additional tables or statistical tests if warranted by the data obtained. The justification for any such additional analyses will be fully documented in the final report.

Descriptive statistics for each of the study endpoints will be provided for the mITT Analysis Set and for both mITT and FT analyses set for the primary endpoint only.

#### 4.1 Disposition of Subjects

Data from subjects who are screened but not treated, subjects in the ITT, mITT, FT analysis sets, as well as study withdrawal data will be summarized using descriptive statistics. This summary will include all subjects screened into the study. The denominator for calculating the percentages will be the set of the ITT.

#### 4.2 Demographics and Baseline Characteristics

Demographic and baseline data as well as disease prognostic factors, medical history and prior medications will be summarized for the ITT analysis set using appropriate descriptive statistics. Baseline characteristics (age, BMI and smoking status) will be presented by categories used for efficacy analyses. Categories for missing data will be presented if necessary. Missing categories will be presented if necessary.

The proportion of subjects who recorded concomitant medications will be tabulated




## 4.3 Compliance

Summary table of compliance data based on Sci-B-Vac injections will be generated for the ITT analysis set.

## 4.4 Primary Endpoint Analysis

The primary endpoint of the study is the Seroprotection rate (SPR), defined as the proportion of subjects with anti-HBs antibody titer at least equal to 10mIU/mI, at Month 7 (i.e. one month after the third immunization with Sci-B-Vac<sup>TM</sup>). In the first Interim Analysis the primary endpoint will be tested on month 4. Subjects early terminated from the study for any reason at any time while having an anti-HBs antibody concentrations  $\geq 10\text{mIU/mI}$  will be considered among those who met endpoint.

The principal analysis of the primary endpoint will employ a non-inferiority analysis [SAS PROC FREQ with binomial (noninf margin=0.09 p=(1- $\alpha$ ) exact)] statement will be used for testing the below hypothesis:

H0: P-p0 ≤ -Margin H1: P-p0 > -Margin

Where p0, the assumed true SPR is 95% and the non-inferiority margin is 9.0%, employing that study will be considered successful if the lower bound of the  $(1-\alpha)$  exact CI will be 86.0% or more.

The rate of responders will be calculated along with 95% confidence interval using Exact binomial method. The final population for statistical analysis will include only subjects who fully comply with the study protocol, have no inclusion/exclusion criteria violation and subjects who early terminated the study but reached the primary endpoint prior to withdrawal (mITT population).

Comparative analysis will be applied for baseline characteristics (such as gender, smoking status, age and BMI) between non seroprotected subjects (i.e. anti-HBsAg antibody<10), seroprotected subjects (ie. anti-HBsAg antibody≥10 mIU/mI) and subjects with Anti-HBs≥100 mIU/mI.

Age categories will be defined by intervals of 5 or 10. BMI will be defined <25 or ≥25. Smoking status will be defined using 5 categories:

Never

Past-smoker;

Light smoker (up to 10 cigs/day)

Moderate smoker (10-19 cigs/day)

Heavy smoker (20 or more cigs/day)BMI categories will be defined <25 and ≥25


## 4.5 Secondary Endpoints Analysis

The secondary endpoints for the study are:

- SPR one month after the first injection and at every month until Month 6 inclusive and at months 9 and 12.
- Percentage of subjects with anti-HBs antibodies titer ≥ 100
- mIU/ml one month after the first injection and then at every month until Month 7 inclusive and at months 9 and 12.
- The geometric mean concentration (GMC) as determined by anti-HBsAg antibody titers at Month 0, then at every month until Month 7 inclusive and at months 9 and 12.

SPR at all time-points as defined above will be analyzed using the principal analysis method as defined for the primary endpoint, and will be presented graphically as well.

The percentage of subjects with anti-HBs antibodies titer ≥ 100 mIU/ml will be calculated from the responders sub-set at each available time-point. Subjects with titer>10 mIU/ml and <100 mIU/ml will be defined 'low-responders'.

The geometric mean concentration (GMC) as determined by anti-HBsAg antibody titers one month after the first injection and at every month until Month 7 inclusive and at months 9 and 12 will be calculated with 95% confidence intervals. Graphical presentation of GMC by month will be generated.

## 4.6 Exploratory Endpoints Analysis

The exploratory endpoints for the study are:

- The anti-preS1 antibody titers measured at Month 0, then at every month until Month 7 inclusive and at months 9 and 12.
- The anti-preS2 antibody titers measured at Month 0, then at every month until Month 7 inclusive and at months 9 and 12.

The geometric mean concentration (GMC) at Month 0, then at every month until Month 7 inclusive and at months 9 and 12 will be displayed across time in order to establish the kinetic of the immunological response during the study.

#### 4.7 Safety analysis

#### 4.7.1 Adverse Events




Adverse events will be recorded from the time when a subject has signed the Informed Consent Form and throughout the study, including the follow-up period. The MedDRA dictionary will be used to standardize the terms used by the investigator to describe the Adverse Events. The following were incorporated into the analyses which will include only Treatment Emergent Adverse Events (TEAEs), namely, events that have started on the day of first study dose or afterwards.

- Summary incidence of adverse events.
- The incidence (no. of subjects) and frequency (no. of events) of TEAEs broken down by System Organ Class (SOC) and by Preferred Term (PT) according to MedDRA dictionary.
- The incidence (no. of subjects) and frequency (no. of events) of TEAEs by SOC, PT and by Severity of event.
- The incidence (no. of subjects) and frequency (no. of events) of TEAEs by SOC, PT and by Relation to study drug.
- The derived dictionary used in the analyses (listing of full glossary).
- Listing of SAEs (regardless if started before or after first study dose) of randomized and dosed subjects captured in the clinical database until database drop date.
- Listing of Non-Treatment Emergent AEs.

#### 4.7.2 Vital Signs

Vital signs will be measured at each treatment visit including at screening and early termination visits whereas unscheduled visit is optional. Analyses of vital signs will be performed in the following manner:

- Descriptive statistics of vital signs before first study dose and afterwards as well as the changes from baseline by scheduled visit will be generated.
- Vital signs will be graded based on table 2 in appendix C of the protocol:





#### **TABLE 2: GRADING OF VITAL SIGNS**

| Vital Signs | Mild<br>(Grade 1) | Moderate<br>(Grade 2) | Severe<br>(Grade 3) | Potentially Life<br>Threatening<br>(Grade 4) |
|---|---|---|---|---|
| Fever (°C)<br>(°F) | 38.0 – 38.4<br>100.4 – 101.1 | 38.5 – 38.9<br>101.2 – 102.0 | 39.0 – 40<br>102.1 – 104 | > 40<br>> 104 |
| Tachycardia - BPM | 101 – 115 | 116 – 130 | > 130 | ER visit or<br>hospitalization for<br>arrhythmia |
| Bradycardia - BPM | 50 – 54 | 45 – 49 | < 45 | ER visit or hospitalization for arrhythmia |
| Hypertension (systolic) -<br>mm Hg | 141 – 150 | 151 – 155 | > 155 | ER visit or hospitalization for malignant hypertension |
| Hypertension (diastolic) -<br>mm Hg | 91 – 95 | 96 – 100 | > 100 | ER visit or<br>hospitalization for<br>malignant hypertension |
| Hypotension (systolic) –<br>mm Hg | 85 – 89 | 80 – 84 | < 80 | ER visit or hospitalization for hypotensive shock |
| Respiratory Rate – breaths per minute | 17 – 20 | 21 – 25 | > 25 | Intubation |

- The incidence (no. of subjects) of vital signs grading will be summarized in a frequency tables.
- Box-Plots of vital signs before first study dose and afterwards by scheduled visit will be provided by request for specific parameters. .

## 4.7.3 Laboratory Test Results

Analyses of safety laboratory data will be performed in the following manner:

- Descriptive statistics of quantitative tests results and changes from baseline by scheduled visit.
- Quantitative laboratory measurements will be categorized with reference to the normal ranges as Low, Normal or High. Incidence tables of laboratory results categories will be presented by visit.
- Incidence tables of CS lab values defined by the PI as well as the individual subject listing will also be provided.
- Box-Plots of laboratory measurements from first study dose and afterwards by scheduled visit will be provided by request for specific parameters.




# 4.7.4 Other Safety Assessments

Summary statistics of other safety evaluations including assessment of ECG, local safety evaluations and pain evaluations (i.e. local reaction grading) will be tabulated and listed.




# 5. APPENDIX I: TABLES TO BE INCLUDED IN THE STATISTICAL REPORT

| Table<br>number | Table Title |
|---|---|
| 14.1 | Demographic and Baseline Data |
| 14.1-1.1<br>14.1-1.2 | Disposition of subjects Primary reason for early discontinuation |
| 14.1-2.1 | Analysis population |
| 14.1-3.1 | Demographic and Baseline data, ITT |
| 14.1-4 | Medical History, ITT |
| 14.1-5 | Baseline Physical Examination, ITT |
| 14.1-6 | Any Concomitant Medication, ITT |
| 14.1-7 | Any Concomitant Non-drug Medication, ITT |
| 14.1.2 | Exposure to Sci-B-Vac injection |
| 14.1.2.1 | Sci-B-Vac injection, ITT |
| 14.2 | Efficacy Analysis |
| 14.2-1 | Seroprotection rate (SPR) by Month, mITT |
| 14.2-2 | Seroprotection rate (SPR) by Month, FT (for first IA mITT who completed month 7 will be presented) |
| 14.2-3 | Secondary Endpoint Analysis: Percentage of Subjects with Anti-HBs≥100 mIU/ml by Month, mITT |
| 14.2-4 | Secondary Endpoint Analysis: Percentage of Subjects with Anti-HBs≥100 mIU/ml) by Month, FT (for first IA mITT who completed month 7 will be presented) |
| 14.2-5 | Geometric means of anti-HBs antibody titers by month, mITT |
| 14.2-6 | Geometric means of anti-HBs antibody titers by month, FT (for first IA mITT who completed month 7 will be presented) |
| 14.2-7 | Frequency of gender by responders (SPR) (at month 4 for first IA) |
| 14.2-8 | Frequency of age categories by responders (SPR) (at month 4 for first IA) |
| 14.2-9 | Frequency of Responders (SPR) by Smoking status and month (month 4 for IA) |
| 14.2-10 | Frequency of Responders (SPR) by BMI categories and month (at month 4 for first IA) |
| 14.2-11 | Geometric means of anti-HBs antibody titers by month and Gender |
| 14.2-12 | Geometric means of anti-HBs antibody titers by month and age categories |
| 14.2-13 | Geometric means of anti-HBs antibody titers by month and Smoking status |
| 14.2-14 | Geometric means of anti-HBsAg antibody titers by month and BMI categories |
| 14.2-15 | Serologic Markers for Hepatits B Infection, ITT |
| 14.3 | Safety Data |
| 14.3.1 | Adverse Events |
| 14.3.1 | Summary Incidence of TEAE (Treatment Emergent Adverse Events), ITT |
| 14.3.1-1 | Summary of Adverse Events by SOC and PT, ITT |





| Table<br>number | Table Title |
|---|---|
| 14.3.1-2 | Summary of Adverse Events by SOC and PT and Severity, ITT |
| 14.3.1-3 | Summary of Adverse Events by SOC and PT and Relation to study drug, ITT |
| 14.3.1-4 | Summary of Serious Adverse Events by SOC and PT, ITT |
| 14.3.2 | Listing of SAEs (if applicable) |
| 14.3.2-1 | Listing of Serious Adverse Events |
| 14.3.4 | Abnormal Laboratory Results |
| 14.3.4-1 | Incidence of Hematology Abnormal Clinically Significant Results |
| 14.3.4-2 | Out of Range Hematology Results |
| 14.3.4-3 | Incidence of Chemistry Abnormal Clinically Significant Results |
| 14.3.4-4 | Out of Range Chemistry Results |
| 14.3.4-5 | Incidence of Urinary Abnormal Clinically Significant Result |
| 14.3.4-6 | Out of Range Urinary Result |
| 14.3.4-7 | Pregnancy test (Females) |
| 14.3.5 | Other Safety Assessment |
| 14.3.5 | Summary statistics of Hematology results by Visit |
| 14.3.6 | Summary statistics of Hematology Changes from Baseline by Visit |
| 14.3.7 | Summary statistics of Chemistry results by Visit |
| 14.3.8 | Summary statistics of Chemistry Changes from Baseline by Visit |
| 14.3.9 | Summary statistics of Urinalysis results by Visit |
| 14.3.10 | Summary statistics of Urinalysis Changes from Baseline by Visit |
| 14.3.11 | Summary of Vital Signs by Visit |
| 14.3.12 | Frequency of Vital Signs Grading by Visit |
| 14.3.13 | Summary of Vital Signs Changes from Baseline (pre-vaccination) by Visit |
| 14.3.14 | ECG Assessment |
| 14.3.15 | Local Reaction |
| 14.3.16 | Any Change in Subject's Health and in concomitant medications since last visit |

Medicine Stat




# 6. APPENDIX II: LISTINGS TO BE INCLUDED IN THE STATISTICAL REPORT

| Listing<br>number<br>16.2<br>16.2.1 | Listing Title Listings by Subject Disposition of Subjects |
|---|---|
| 16.2.1-1 | Disposition of subjects, ITT |
| 16.2.4 | Demographic, baseline and Medical History data |
| 16.2.4-1 | Demographic and baseline data |
| 16.2.4-2 | Medical History |
| 16.2.4-2a | Reported Medical History for Screening Failures Baseline Physical Examination |
| 16.2.4-3<br>16.2.4-4 | Concomitant Medications |
| 16.2.4-4 | Concomitant Medications Concomitant Non-drug Treatments |
| 16.2.4-6.1 | Serology Markers for Hepatitis B Infection at Screening/ Visit 11/ET |
| 16.2.4-6.2 | Early Serology Markers for Hepatitis B Infection monitored during the study |
| 16.2.5 | Exposure to Sci-B-Vac Injection |
| 16.2.5-1 | Compliance data |
| 16.2.6 | Individual Efficacy response data |
| 16.2.6-1 | Serologic Response to Immunization |
| 16.2.7 | Adverse event listings |
| 16.2.7-1 | Treatment Emergent Adverse Events |
| 16.2.7-2 | Non-Treatment Emergent Adverse Events |
| 16.2.7-3 | Full Glossary of Adverse Events |
| 16.2.8 | Listing of individual laboratory and other assessments by subject |
| 16.2.8-1 | Abnormal Clinically Significant Hematology Results |
| 16.2.8-2 | Hematology Results |
| 16.2.8-3 | Abnormal Clinically Significant Chemistry Results |
| 16.2.8-4<br>16.2.8-5 | Chemistry Results |
| 16.2.8-6 | Abnormal Clinically Significant Urinalysis Results |
| 16.2.8-7-1 | Urinalysis Results Test for Pregnancy (Females) |
| 16.2.8-7-1 | Previous pregnancies data for subject S1168 |
| 16.2.8-7.3 | Current pregnancy data for subject S1168 |
| 16.2.8-8 | Vital Signs |
| 16.2.8-9 | ECG Assessment |
| 16.2.8-10 | Local Reaction grading |
| 16.2.8-11 | Any Change in subject's health and in concomitant medications since last |
| | visit |
| 16.4 | Eligibility |
| 16.4-1 | Inclusion/ Exclusion Criteria |




| Listing<br>number | Listing<br>Title |
|-------------------|-------------------------|
| 16.4.2 | Visit dates |
| 16.4.2-1 | Visit dates per Subject |
| 16.4.4-1 | Protocol deviations |

## 7. APPENDIX III: FIGURES

| Figure<br>number | Title |
|---|---|
| Figure 1 | SPR by month, mITT |
| Figure 2 | SPR by month, FT (for first IA mITT who completed Month 7) |
| Figure 2.1 | Percentage of non-responder, responder and high-responder to Sci-B-Vac <sup>™</sup> by Month, mITT (second interim analysis) |
| Figure 3 | Geometric Mean of anti-HBs Antibody titers by month, mITT |
| Figure 4 | Geometric Mean of anti-HBs Antibody titers by month, FT (for first IA mITT who completed Month 7) |
| Figure 5 | Geometric Mean of anti-HBs Antibody titers by month and Gender |
| Figure 6 | Geometric Mean of anti-HBs Antibody titers by month and Age |
| Figure 7 | Geometric Mean of anti-HBs Antibody titers by month and Smoking status |
| Figure 8 | Geometric Mean of anti-HBs Antibody titers by month and BMI |

<sup>\*</sup> Box plots for laboratory results and vital signs will be generated for specific parameters, based on the results and the sponsor's request.







# 8. APPENDIX IV: LISTINGS OF SCREENING FAILURES

| Listing<br>number | Listing Title |
|---|---|
| 18.1 | Demographic and Baseline data |
| 18.2.4-1 | Demographic and baseline data |
| 18.2.4-2 | Medical History |
| 18.2.4-3 | Baseline Physical Examination |
| 18.2.4-6 | Baseline Serology Markers for Hepatitis B Infection |
| 18.2.5 | Reasons for Screening Failure |
| 18.2.5 | Reasons for Screening Failure |
| Table | Summary of Reasons for Screening Failure |
| 18.2.5 | |
| 18.2.8 | Listing of individual laboratory and other assessments by subject |
| 18.2.8-2 | Hematology Results |
| 18.2.8-4 | Chemistry Results |
| 18.2.8-6 | Urinalysis Results |
| 18.2.8-7 | Pregnancy Blood Test (Females) |
| 18.2.8-8 | Vital Signs |
| 18.2.8-9 | ECG Assessment |
| 18.2.8-10 | Screening Serology |





# 9. VERSION HISTORY:

| Version | Date | Section | Changes | Done By |
|---|---|---|---|---|
| 1.0 | 22/Feb/2016 | | Original Release | |
| 1.1 | 23/Jun/2016 | abbreviati<br>ons | Added/deleted abbreviations | Daphna<br>Goffer/ |
| | | 2.3 | Study flow chart was revised according to changes in the protocol | Nathalie<br>Machluf |
| | | | Added analyses by gender, age, BMI and smoking, | |
| 2.0 | 23/Jul/2016 | 4.4 | Defining age, BMI and smoking categories | |
| | | | Adding figures for SPR, GMC | Daphna |
| | | 4.5 | Delete GMC ratio | Goffer/<br>Nathalie |
| | | 2.7 | Update interim analysis report description | Machluf |
| 3.0 | 18/Sep/2016 | Appendix<br>I and II | Minor edits to tables and listings names/tables | Daphna<br>Goffer/<br>Nathalie |
| | | 4.7.2 | Add text to table 2 (vital signs grading) | Machluf |
| 4.0 | 24/May/2017 | 2.7 | Adding second Interim Analysis | |
| | | Appendix<br>I and III | Minor edits to tables names | - |
| | | Appendix<br>II | Correct order of listings Add listings 16.2.8-7-2 and 16.2.8-7-3 | Daphna<br>Goffer |
| | | 11 | Add listings 10.2.0-7-2 and 10.2.0-7-3 | Gonei |




#### 10. APPROVAL FOR IMPLEMENTATION OF

## **Statistical Analysis Plan**

Title: AN OPEN LABEL, SINGLE ARM, SINGLE

CENTER CLINICAL STUDY IN HEALTHY
SUBJECTS TO QUALIFY AN IN-HOUSE

REFERENCE STANDARD BATCH OF SCI-B-

**VAC**<sup>TM</sup>

Reference: SciB018 SAP

Version: V4.0

Date effective: 25-May-2017

Author: Daphna Goffer Statistician, Medistat

Author's signature: Date: 25 May 2017

Reviewed By: Gil Harari, CEO Statistician, Medistat

Reviewer's Date: 25 May 2017

signature:






The above Statistical Analysis Plan has been reviewed and approved by the Sponsor:

Name of Approver: Nathalie Machluf

Position: Director Clinical and Regulatory Affairs

Signature: Date: 25/5/2017